CLINICAL TRIAL: NCT01120340
Title: Evaluation of Efficacy of Mesalamine in the Long-term Prevention of Diverticulitis Flares
Acronym: DIV-01/04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Sofar
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Diverticular Disease
MeSH Terms: conditions — Diverticular Diseases | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mesalamine (Active Comparator): Posology: mesalamine: 1,6 g/die for ten days every month for 24 months
  Interventions: Drug: mesalamine
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: mesalamine — mesalamine: 1.6 g/die for ten days/month until 24 months
  Arms: mesalamine
Other: placebo — 2 pills/day for ten days/month until 24 months
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether mesalamine is effective vs. placebo in the prevention of diverticulitis flares in a 24-months follow-up.

The primary end-point of the study is the incidence of diverticulitis flares. Will be made a clinical diagnosis of uncomplicated diverticulitis: fever, leukocytosis, abdominal pain and altered intestinal motility.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* both males and females patients
* positive history of acute diverticulitis flare during the last year. The patients will be recruited only after the complete clinical remission of diverticulitis flare.
* patients who have given their free and informed consent

Exclusion Criteria:

* complicated diverticulitis(fistulas, stenosis, abscesses and/or bleeding)
* ascertained hypersensitivity to the salicylates
* any severe pathology that can interfere with the treatment or the clinical or instrumental test of the trial
* clinically significant renal or hepatic impairment
* esophageal, gastric or duodenal ulcer within 30 days prior to randomisation
* patients with active malignancy of any type, or history of a malignancy (patients with a history of malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrollment are also acceptable)
* treatment with any investigational drug within the previous 30 days
* treatment with lactulose or with any compound that lowering the colonic pH can prevent the release of the active moiety from the tablets
* recent history or suspicion of alcohol abuse or drug addiction
* patients who become unable to conform to protocol
* patients with ascertained pregnancy
* previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
diverticulitis relapse | 24 months

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - Ospedale di Seriate, Seriate, Bergamo
  - Ospedale di Esine, Esine, Brescia
  - Ospedale Maggiore, Crema, Cremona
  - Ospedale di Desio, Desio, Milano
  - Ospedale di Garbagnate M.se, Garbagnate Milanese, Milano
  - Ospedale C. Borella, Giussano, Milano
  - Ospedale Civile, Legnano, Milano
  - A.O. G. Salvini, Rho (MI), Milano
  - Policlinico di Monza, Monza, Monza-Brianza
  - Ospedale S. Antonio Abate, Gallarate, Varese
  - Azienda ULSS, Belluno
  - Poliambulanza, Brescia
  - Ospedale A. Manzoni, Lecco
  - Ospedale G. Bosco, Torino
  - Ospedale Maria Vittoria, Torino
  - Ospedale Molinette, Torino
  - Ospedale S. Chiara, Trento

REFERENCES:
- [Derived] Parente F, Bargiggia S, Prada A, Bortoli A, Giacosa A, Germana B, Ferrari A, Casella G, De Pretis G, Miori G; "Gismi Study Group". Intermittent treatment with mesalazine in the prevention of diverticulitis recurrence: a randomised multicentre pilot double-blind placebo-controlled study of 24-month duration. Int J Colorectal Dis. 2013 Oct;28(10):1423-31. doi: 10.1007/s00384-013-1722-9. Epub 2013 Jun 12. PMID 23754545